CLINICAL TRIAL: NCT02076282
Title: MRI for Radiotherapy Treatment Planning of Stage III NSCLC: an MRI Optimization Study in Healthy Volunteers and Patients
Brief Title: MRI Optimization Study in Stage III NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, M. van Vulpen, MD, PhD, UMC Utrecht
Other Study IDs: NL46711.041.13
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Stage III Non-small Cell Lung Cancer
Keywords: Stage III non-small cell lung cancer; Optimization; MRI; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy volunteers 1 MRI scan: Healthy volunteers, recruited at the UMC Utrecht, older than 18, who do not meet the exclusion criteria of the department of Radiology.
  Healthy volunteers will receive 1 MRI scan without contrast agent.
  Interventions: Other: 1 MRI scan
- Patients with stage III NSCLC, 1 MRI scan: Patients with histopathologically or cytologically proven stage III NSCLC (excluding T4N0), older than 18, with a recent (≤ 21 days) GFR value available
  Patients will receive 1 MRI scan with contrast agent.
  Interventions: Other: 1 MRI scan

INTERVENTIONS:
Other: 1 MRI scan — For healthy volunteers: 1 MRI scan without contrast
  For patients: 1 MRI scan with contrast

SUMMARY:
Radiation therapy uses radiation to treat lung tumors and metastases in the mediastinum. In order to irradiate as precise as possible, and in order to evaluate the effect of radiation treatment, it is important to depict the lung tumor and the lymph node metastases as accurate as possible. Currently, radiation oncologists use PET-CT for this purpose. However, PET-CT does have its drawbacks, and partly because of this, large volumes are irradiated in current treatment.

The investigators believe that MRI can be used to improve depiction of the tumor and lymph nodes and of their motion. However, there is currently no MRI protocol available which is aimed at improving radiotherapy.

In this study, the investigators want to select the optimal MRI settings for depiction of the lung tumor, the lymph node metastases and their movement.

The investigators plan to do this by first examining 10 healthy volunteers, followed by 20 patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
Rationale:

- Patients with stage III non-small cell lung cancer (NSCLC) have a poor survival due to inadequate loco-regional control. Increasing the dose will lead to better loco-regional control and survival. However, with the current treatment planning strategies, increasing this dose would result in intolerable toxicity of the organs at risk (OARs, healthy tissue surrounding the tumor). Therefore, new treatment planning strategies have to be developed to improve local control and therefore overall survival of patients with stage III NSCLC.

Currently, the radiation oncologist uses a combination of imaging modalities for the delineation of the lung tumor and lymph nodes: four-dimensional (4D)- computed tomography (CT) scan, CT-scan with intravenous contrast and the positron emission tomography (PET)-CT with fluorodeoxyglucose as a radioactive tracer. However these imaging modalities have some disadvantages.In current clinical practice, large treatment volumes are irradiated. This results in an increased dose to OARs. Consequently, further increasing of the dose to the tumor would result in intolerable toxicity.

The investigators believe that MRI can be used to improve visualization of the tumor and lymph nodes and characterize their motion, based on promising results in recent literature. MRI can potentially be used to obtain more accurate (thus smaller) treatment volumes. This will lead to a smaller dose to the OARs and enable safe dose escalation.

Unfortunately there are no MRI protocols in the literature available aimed at radiotherapy of lung cancer.

The objective of this study is twofold. The investigators would first like to use MRI in volunteers to select the appropriate techniques for motion compensation. Furthermore, MRI settings will be sought which can be used to image lung and mediastinal parenchyma.

Second, the investigators would like to assess the MRI sequences found in volunteers for the visualization of tumors and lymph nodes in patients with stage III NSCLC. Furthermore, the investigators would like to assess if MRI can be used for (automatic) motion characterization of tumor, lymph nodes and organs at risk.

The sequences found in this study will be used in a future study on the added value of MRI for radiotherapy treatment planning of stage III NSCLC, in which MRI will also be compared to PET-CT.

Objectives:

* To select the appropriate techniques to image lung and mediastinal parenchyma. Furthermore, MRI settings will be sought which can be used for motion compensation.
* To optimize and validate MRI for the visualization and motion characterization of tumor, lymph nodes and mediastinal parenchyma in patients with stage III NSCLC.

Study design: Observational study.

Study population:10 healthy volunteers and 20 patients with pathologically proven stage III NSCLC with lymph node metastases (i.e. excluding T4N0) referred to the department of Radiation Oncology.

Procedure: Healthy volunteers will undergo an MRI scan without intravenous contrast. Patients will undergo a contrast-enhanced MRI scan.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

* Healthy volunteers will undergo an MRI scan with a maximal duration of 45 minutes. One visit to the hospital (lasting approximately 75 minutes) is required and the healthy volunteers will receive a gift voucher with a value of 25 euros. MRI-safety screening is required before the MRI scan, and consists of routine screening according to the clinical guidelines as determined by the Department of Radiology of the UMCU.
* Patients will undergo an MRI scan with a maximal duration of 45 minutes. The total visit to the department (including patient preparation, changing of clothes etc.) will last approximately 75 minutes. For determination of renal function, a recent value of the Glomerular Filtration Rate (GFR) (≤21 days) has to be available.

After proper screening, the use of MRI is safe. The use of gadolinium contrast (Gadovist) has a very low risk of contrast induced allergy. For the patients included in the study there is no individual benefit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

  1. ≥18 years.
  2. Written informed consent
* Patients

  1. Patients with histopathologically or cytologically proven stage III NSCLC (excluding T4N0) referred to the department of Radiation Oncology
  2. ≥ 18 years.
  3. Written informed consent.
  4. Recent (≤ 21 days) GFR value available

Exclusion Criteria:

* Healthy volunteers:

  1. Volunteers who meet exclusion criteria for MRI following the protocol of the department of Radiology of the UMC Utrecht
* Patients:

  1. Patients who meet exclusion criteria for MRI following the protocol of the department of Radiology of the UMC Utrecht.
  2. Patients for whom lying still in a supine position for 45 minutes is physically too strenuous (e.g. due to orthopnea).
  3. Glomerular Filtration Rate (GFR) of <30 mL/min/1.73m2 (UMCU protocol 'MRI Contra-indicaties', Version 3 January 2013).
  4. Patients with nephrogenic systemic fibrosis, nephrogenic fibrosing dermopathy or severe renal insufficiency (UMCU protocol 'MRI Contra-indicaties', Version 3 January 2013).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 10 healthy volunteers
  * 20 patients with pathologically proven stage III NSCLC with lymph node metastases (i.e. excluding T4N0) referred to the department of Radiation Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Optimization and validation of an MRI scanning protocol | Healthy volunteers: 1 time point, patients: at start of radiation treatment
  The aim of this study is to optimize and validate an MRI scanning protocol for patients with stage III NSCLC aimed at radiotherapy purposes (i.e. tumor delineation and motion characterization).Optimization is defined by the quality of the images.
  In healthy volunteers, the study endpoint is to select the sequences with the highest quality.
  Quality of the scans will be assessed by rating the motion artifacts and visibility of the lung and mediastinal parenchyma. This will be done by a group of experts (radiologist, radiation oncologist, medical physicist, MRI physicist and a researcher).
  The sequences with the highest quality will be optimized in patients. In patients, the quality will be assessed by rating of the images on the following criteria:
  * Contrast between tumor/lymph nodes and their surrounding tissue.
  * Depiction of tumor, lymph node and mediastinal organ motion.
  * Presence of artifacts.

SECONDARY OUTCOMES:
Power analysis | Healthy volunteers: one time point, patients: start of radiation therapy
  The results of this optimization study will be used for the power analysis of consecutive studies.

CONTACTS AND LOCATIONS:
Overall Officials: Marco van Vulpen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center, Utrecht, Utrecht, Netherlands